CLINICAL TRIAL: NCT03025087
Title: Hydroxychloroquine and Cognitive Function After Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Showed no benefit
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00046611
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Results first posted 2024-06-12 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Individuals Undergoing Cardiac and General Surgery
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase 1 (Experimental): 6 evaluable subjects (3 cardiac, 3 noncardiac patients): 1000 mg HCQ on the day prior to surgery.
  Interventions: Drug: Hydroxychloroquine
- Phase 2 (Experimental): 6 evaluable subjects (3 cardiac, 3 noncardiac patients): 1000 mg HCQ on the day prior to surgery followed by 400 mg daily until the day of MRI imaging on postoperative day 1-5
  Interventions: Drug: Hydroxychloroquine
- Phase 3 (Experimental): 6 evaluable cardiac subjects 1000 mg HCQ on the day prior to surgery followed by 400 mg twice daily (800 mg total) until the day of MRI imaging on postoperative day 1-5.
  Interventions: Drug: Hydroxychloroquine
- Phase 4 (Experimental): 6 evaluable cardiac subjects: 1000 mg HCQ on the day prior to surgery followed by 500 mg twice daily (1000 mg total) until the day of MRI imaging on postoperative day 1-5.
  Interventions: Drug: Hydroxychloroquine
- Phase 5 (Experimental): 6 evaluable cardiac subjects: 1000 mg HCQ 1-2 hours after separation from CPB followed by the highest tolerated dose from the previous 4 phases divided into 2 equal daily doses until the day of MRI imaging on postoperative day 1-5.
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Participants will be getting hydroxychloroquine

SUMMARY:
The purpose of this study is to determine whether hydroxychloroquine decreases the relative leakage of the brain barrier after surgery.

DETAILED DESCRIPTION:
Hydroxychloroquine will be administered preoperatively to 30 patients undergoing cardiac surgery. All patients will undergo magnetic resonance imaging (MRI) with gadolinium in the post-operative period before hospital discharge in order to assess blood-brain barrier permeability.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 50 years old.
2. Patients scheduled to undergo cardiac surgery (CABG, CABG + Valve, Valve) with CPB.
3. Patient has voluntarily signed and dated the study-specific informed consent form approved by Duke University Health System Institutional Review Board (DUHS IRB)

Exclusion Criteria:

1. Cardiac surgery scheduled to be performed without cardiopulmonary bypass
2. Patients requiring emergent operation
3. Patients with a history of myocardial infarction within 7 days of surgery
4. Patients with a history of porphyria, psoriasis, chronic dermatitis, or retinal disease
5. Patients receiving preoperative digoxin
6. Patients with symptomatic cerebrovascular disease with substantial residual deficit
7. Patients with a history of alcohol abuse within 2 years of screening
8. Patients with a history of psychiatric illness and/or anxiety requiring medical treatment.
9. Patients with impaired liver and/or kidney functions (AST, ALT 2 times the upper limit of normal)
10. Patients with impaired renal functions (GFR < 30ml/min)
11. Patients with less than a 7th-grade education or unable to read and thus unable complete the neuropsychological testing
12. Patients scoring < 26 on a baseline Mini Mental State examination (MMSE) or scoring >27 on the Center for Epidemiological Studies - Depression (CES-D) scale
13. Female subjects of childbearing potential who have had menstrual period within the past two years
14. Patients with bodily implants unsafe for MRI use
15. Patients with a history of claustrophobia
16. Known or suspected hypersensitivity to quinine (chloroquine or hydroxychloroquine)
17. Patient with pre-existing diagnosis of G6PD deficiency
18. Patients who have participated in another interventional clinical study within the previous 30 days
19. Any other concurrent disease or illness that, in the opinion of the investigator, makes the patient unsuitable for the study
20. Major ophthalmologic comorbidities (ex: ruptured globe, retinal vascular occlusive disease, retinal artery occlusion, anterior ischemic optic neuropathy, media opacification due to corneal abnormalities or cataract that prevent ocular and optical coherence tomography examination, glaucoma, age-related macular degeneration, history of intravitreal injections, and macular edema)
21. Patients who have received chemotherapy in the last 12 months
22. Patient with a QTc of 450 msec or greater (or 500 msec or greater in those with known IVCD, RBBB, or LBBB) at baseline will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Mathew, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Health, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing cardiac or noncardiac surgery were recruited at Duke University Medical Center.
Pre-assignment Details: There was no enrollment in Phase 3, Phase 4, or Phase 5.
Period: Overall Study
Arm/Group | Phase 1 | Phase 2 | Phase 3 | Phase 4 | Phase 5
Started | 12 | 12 | 0 | 0 | 0
Completed | 6 | 6 | 0 | 0 | 0
Not Completed | 6 | 6 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Not completed — Unable to complete MRI | 2 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data not collected on eight participants. There was no enrollment in Phase 3, Phase 4, or Phase 5.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 | Phase 3 | Phase 4 | Phase 5 | Total
Number analyzed (Participants) | 8 | 8 | 0 | 0 | 0 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (4.5) | 64.8 (5.8) |  |  |  | 64.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 |  |  |  | 6
  Male | 6 | 4 |  |  |  | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  |  |  | 0
  Not Hispanic or Latino | 8 | 8 |  |  |  | 16
  Unknown or Not Reported | 0 | 0 |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  |  | 0
  Asian | 0 | 1 |  |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  | 0
  Black or African American | 0 | 0 |  |  |  | 0
  White | 8 | 7 |  |  |  | 15
  More than one race | 0 | 0 |  |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 |  |  |  | 16

OUTCOME MEASURES:

1. Primary Outcome: Ktrans Volume Transfer Constant
Description: Ktrans represents the "permeability" or "leakage" constant across the blood-brain barrier and is calculated by measuring the amount of gadolinium-based contrast agent in the extravascular-extracellular space. Ktrans is a constant assessed on the postoperative MRI and has no units of measure.
Time Frame: Postoperative day 1-5
Population: Participants who completed the MRI.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 4 | 4
unitless | 0.225 (0.108) | 0.418 (0.069)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: No enrollment in Phase 3, Phase 4, or Phase 5.
Arm/Group | Phase 1 | Phase 2 | Phase 3 | Phase 4 | Phase 5
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/12 | 3/12 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=12) | Phase 2 (N=12) | Phase 3 (N=0) | Phase 4 (N=0) | Phase 5 (N=0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=12) | Phase 2 (N=12) | Phase 3 (N=0) | Phase 4 (N=0) | Phase 5 (N=0)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT03025087/Prot_SAP_000.pdf